CLINICAL TRIAL: NCT02740205
Title: Efficacy and Safety of the Implementation of an Algorithm for Enteral Nutrition Support Compared With Traditional Practice in Non-critical Patients: Randomized Clinical Trial, Simple Blind.
Brief Title: Efficacy and Safety of the Implementation of an Algorithm for Enteral Nutrition Support.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Aurora Elizabeth Serralde Zúñiga, MD, PhD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1390
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Malnutrition
Keywords: Patients with Enteral Feeding
MeSH Terms: conditions — Malnutrition | interventions — Algorithms; Clinical Protocols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Hospital's standard EN support at the discretion of the Clinical Nutrition Service that is composed by physicians, dietitians, and students, provides nutritional assessments, recommendations and consultations for the in-patients that required nutrition support during their hospitalization stay. There is no protocols or algorithms for the nutritional support in our institution, the currently clinical practice of the EN is prescribed by the physician, dietitians and students during the morning rounds each 24h, the kind of EN formulas prescribed depends of the clinical status of the patient, when the patients required protein supplements modular protein supplements are added.
- Algorithm for enteral nutrition support (Experimental): Initial infusion of 20 to 40 ml/h, evaluated the tolerability in the next 8-12h, then the infusion can be increased 25 ml/ 8-12h for gastric infusion and 10-20 ml/h for the post-pyloric feeding, for bolus infusion an initial infusion of 125 ml each 4-5hrs and evaluated the tolerability in the next 8-12h. If the subject present intolerability to the EN, the action in the algorithm indicate hold the infusion 4h then restarted at 10 ml/h with prokinetics agents rather than the suspension. As a part of the intervention, several educational sessions for the medical, nutritionist and nurse staff were performed during the period of the study.
  Interventions: Other: Algorithm for enteral nutrition support

INTERVENTIONS:
Other: Algorithm for enteral nutrition support — Enteral nutrition support prescribed by the Clinical Nutrition Service under the instructions of the algorithm based on evidence
  Other Names: Protocol for enteral nutrition support
  Arms: Algorithm for enteral nutrition support

SUMMARY:
The purpose of this trial is to evaluate the efficacy and safety of the implementation of an Algorithm for enteral nutrition support compared with usual standard practice in non-critical hospitalized patients: ASNET algorithm.

DETAILED DESCRIPTION:
The algorithms for the enteral nutrition support also called protocols had been developed and implemented in the intensive care units (ICU) across the world to enhance the provision of calories and proteins via enteral nutrition (EN), increasing the proportion of patients that received an optimal amount (80-85% of their energy and protein requirements), and decreasing the caloric and protein debt. The algorithm includes different designs and interventions, the variability of the design is because the algorithm is adapted to the local necessities.

The principal reason for the algorithm implementation is the rate of underfed (receiving <80% of prescribed of energy and protein requirements) as a result of numerous causes 26% considered avoidable events, and the variation of the clinical practice. There's a universal consensus that the EN is the principal artificial way for the macro-micro nutrients delivery, it comes with the novelty "if the gut works, use it or prepare to lose it". The evidence shows that the EN is more physiological and when the patients received the optimal amount of EN the clinical outcomes (length of hospital stay, mortality and infection rates) can decrease significantly. In average 74% of the patients in the ICU that received EN are underfed, in Mexico 71% of the hospitalized patients with EN in non-critical areas are underfed, receiving only 61% of their energy requirements during their hospitalization.

The investigators propose an algorithm for the EN support based on evidence, in order to avoid the variability in the prescription that include a prediction equation according to the BMI to calculate the energy and protein requirements. The algorithm propose the range for the initial infusion for the gastric and post-pyloric feeding in continuous infusion and evaluated the tolerability, if there is no signs and symptoms of intolerance then the infusion can be increased. If the subject present intolerability to the EN (diarrhea, abdominal distention), an action in the algorithm indicate options rather than the suspension. Moreover when the EN is interrupt for a reason that is not intolerance and only if the patient already reach the goal rate the compensatory feed table can be use it. As a part of the intervention, several educational sessions for the medical, nutritionist and nurse staff were performed during the period of the study.

The investigators hypothesize that the implementation of the algorithm for EN support will increase the amount of energy and protein safely and effectively to the patients compared with the usual practice.

The purpose of this study is to evaluate the efficacy and safety of the implementation of an algorithm for EN support (ASNET).

ELIGIBILITY:
Inclusion Criteria:

* Candidate to receive exclusively enteral nutrition
* Consent form signed

Exclusion Criteria:

* Patients in critical areas
* Carcinomatosis
* ICU admission
* Intestinal failure
* Receiving tube feeding prior to hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2020-08-13 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Adequacy of enteral nutrition | 4 days
  The percentage of energy and proteins received by the patient trough tube feeds in contrast with the prescription

SECONDARY OUTCOMES:
Security variable | 30 days
  The rate of gastrointestinal complications:
  diarrhea (>500cc), abdominal distention, emesis.

CONTACTS AND LOCATIONS:
Overall Officials: Aurora E Serralde-Zúñiga, MD,PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mackenzie SL, Zygun DA, Whitmore BL, Doig CJ, Hameed SM. Implementation of a nutrition support protocol increases the proportion of mechanically ventilated patients reaching enteral nutrition targets in the adult intensive care unit. JPEN J Parenter Enteral Nutr. 2005 Mar-Apr;29(2):74-80. doi: 10.1177/014860710502900274. PMID 15772383
- [Background] Kiss CM, Byham-Gray L, Denmark R, Loetscher R, Brody RA. The impact of implementation of a nutrition support algorithm on nutrition care outcomes in an intensive care unit. Nutr Clin Pract. 2012 Dec;27(6):793-801. doi: 10.1177/0884533612457178. PMID 23135707
- [Background] Arabi Y, Haddad S, Sakkijha M, Al Shimemeri A. The impact of implementing an enteral tube feeding protocol on caloric and protein delivery in intensive care unit patients. Nutr Clin Pract. 2004 Oct;19(5):523-30. doi: 10.1177/0115426504019005523. PMID 16215149
- [Background] Heyland DK, Cahill NE, Dhaliwal R, Wang M, Day AG, Alenzi A, Aris F, Muscedere J, Drover JW, McClave SA. Enhanced protein-energy provision via the enteral route in critically ill patients: a single center feasibility trial of the PEP uP protocol. Crit Care. 2010;14(2):R78. doi: 10.1186/cc8991. Epub 2010 Apr 29. PMID 20429886
- [Background] Ventura AM, Waitzberg DL. Enteral nutrition protocols for critically ill patients: are they necessary? Nutr Clin Pract. 2015 Jun;30(3):351-62. doi: 10.1177/0884533614547765. Epub 2014 Sep 23. PMID 25249598
- [Background] Martin CM, Doig GS, Heyland DK, Morrison T, Sibbald WJ; Southwestern Ontario Critical Care Research Network. Multicentre, cluster-randomized clinical trial of algorithms for critical-care enteral and parenteral therapy (ACCEPT). CMAJ. 2004 Jan 20;170(2):197-204. PMID 14734433
- [Background] Heyland DK, Cahill N, Day AG. Optimal amount of calories for critically ill patients: depends on how you slice the cake! Crit Care Med. 2011 Dec;39(12):2619-26. doi: 10.1097/CCM.0b013e318226641d. PMID 21705881
- [Background] Taylor B, Brody R, Denmark R, Southard R, Byham-Gray L. Improving enteral delivery through the adoption of the "Feed Early Enteral Diet adequately for Maximum Effect (FEED ME)" protocol in a surgical trauma ICU: a quality improvement review. Nutr Clin Pract. 2014 Oct;29(5):639-48. doi: 10.1177/0884533614539705. PMID 25155862
- [Background] Bowman A, Greiner JE, Doerschug KC, Little SB, Bombei CL, Comried LM. Implementation of an evidence-based feeding protocol and aspiration risk reduction algorithm. Crit Care Nurs Q. 2005 Oct-Dec;28(4):324-33; quiz 334-5. doi: 10.1097/00002727-200510000-00004. PMID 16239821
- [Background] Woien H, Bjork IT. Nutrition of the critically ill patient and effects of implementing a nutritional support algorithm in ICU. J Clin Nurs. 2006 Feb;15(2):168-77. doi: 10.1111/j.1365-2702.2006.01262.x. PMID 16422734
- [Background] Martins JR, Shiroma GM, Horie LM, Logullo L, Silva Mde L, Waitzberg DL. Factors leading to discrepancies between prescription and intake of enteral nutrition therapy in hospitalized patients. Nutrition. 2012 Sep;28(9):864-7. doi: 10.1016/j.nut.2011.07.025. Epub 2011 Nov 25. PMID 22119484
- [Background] Lottes Stewart M. Nutrition support protocols and their influence on the delivery of enteral nutrition: a systematic review. Worldviews Evid Based Nurs. 2014 Jun;11(3):194-9. doi: 10.1111/wvn.12036. Epub 2014 May 19. PMID 24841717
- [Background] Cahill NE, Murch L, Cook D, Heyland DK; Canadian Critical Care Trials Group. Improving the provision of enteral nutrition in the intensive care unit: a description of a multifaceted intervention tailored to overcome local barriers. Nutr Clin Pract. 2014 Feb;29(1):110-7. doi: 10.1177/0884533613516512. Epub 2013 Dec 16. PMID 24344255
- [Background] Peev MP, Yeh DD, Quraishi SA, Osler P, Chang Y, Gillis E, Albano CE, Darak S, Velmahos GC. Causes and consequences of interrupted enteral nutrition: a prospective observational study in critically ill surgical patients. JPEN J Parenter Enteral Nutr. 2015 Jan;39(1):21-7. doi: 10.1177/0148607114526887. Epub 2014 Apr 7. PMID 24714361
- [Background] Heyland DK, Cahill NE, Dhaliwal R, Sun X, Day AG, McClave SA. Impact of enteral feeding protocols on enteral nutrition delivery: results of a multicenter observational study. JPEN J Parenter Enteral Nutr. 2010 Nov-Dec;34(6):675-84. doi: 10.1177/0148607110364843. PMID 21097768
- [Background] Langkamp-Henken B. If the gut works, use it: but what if you can't? Nutr Clin Pract. 2003 Dec;18(6):449-50. doi: 10.1177/0115426503018006449. No abstract available. PMID 16215080
- [Background] Barr J, Hecht M, Flavin KE, Khorana A, Gould MK. Outcomes in critically ill patients before and after the implementation of an evidence-based nutritional management protocol. Chest. 2004 Apr;125(4):1446-57. doi: 10.1378/chest.125.4.1446. PMID 15078758
- [Background] Braunschweig CL, Levy P, Sheean PM, Wang X. Enteral compared with parenteral nutrition: a meta-analysis. Am J Clin Nutr. 2001 Oct;74(4):534-42. doi: 10.1093/ajcn/74.4.534. PMID 11566654
- [Background] Heyland DK, Dhaliwal R, Wang M, Day AG. The prevalence of iatrogenic underfeeding in the nutritionally 'at-risk' critically ill patient: Results of an international, multicenter, prospective study. Clin Nutr. 2015 Aug;34(4):659-66. doi: 10.1016/j.clnu.2014.07.008. Epub 2014 Jul 19. PMID 25086472
- [Background] Baca Molina GP, Pena Corona M. [Prevalence of enteral patients with suboptimal feeding at Centro Medico Lic. Adolfo Lopez Mateos]. Nutr Hosp. 2015 Apr 1;31(4):1597-602. doi: 10.3305/nh.2015.31.4.8353. Spanish. PMID 25795946
- [Background] MacLaren R. Intolerance to intragastric enteral nutrition in critically ill patients: complications and management. Pharmacotherapy. 2000 Dec;20(12):1486-98. doi: 10.1592/phco.20.19.1486.34853. PMID 11130221
- [Background] Kim H, Stotts NA, Froelicher ES, Engler MM, Porter C. Why patients in critical care do not receive adequate enteral nutrition? A review of the literature. J Crit Care. 2012 Dec;27(6):702-13. doi: 10.1016/j.jcrc.2012.07.019. Epub 2012 Oct 17. PMID 23084129
- [Derived] Ortiz-Reyes LA, Castillo-Martinez L, Lupian-Angulo AI, Yeh DD, Rocha-Gonzalez HI, Serralde-Zuniga AE. Increased Efficacy and Safety of Enteral Nutrition Support with a Protocol (ASNET) in Noncritical Patients: A Randomized Controlled Trial. J Acad Nutr Diet. 2018 Jan;118(1):52-61. doi: 10.1016/j.jand.2017.09.020. PMID 29274643